CLINICAL TRIAL: NCT01510015
Title: Evaluation of the Effects of Psychological and Pharmacological Treatment of Psycho-stimulant and Cannabis-dependent Users in Kfar Izun in Israel
Brief Title: Evaluation of the Effects of Treatment of Psycho-stimulant and Cannabis-dependent Users in Israel
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, Michal Roll PhD,MBA, Head of Research and Development, Tel-Aviv Sourasky Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0503-11-TLV
Record Dates: First submitted 2011-12-27; First posted 2012-01-13 (Estimated); Last update posted 2012-01-13 (Estimated); Status verified 2012-01

CONDITIONS: Cannabis Dependence; Psychostimulant Dependence
Keywords: cannabis; psychostimulants; psychosis
MeSH Terms: conditions — Marijuana Abuse; Psychotic Disorders | interventions — Risperidone; Psychotherapy, Group

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anti-psychotic medication (Active Comparator): Participants are treated with psychological treatment both group and individually as well as medications according to their mental condition.
  Interventions: Drug: Risperidone
- Counseling (Active Comparator): Participants will receive individual and group therapy
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Risperidone — variable dose
  Other Names: Individual and group therapy

SUMMARY:
This study evaluates the effects of psychological and pharmacological treatment of regular users of cannabis and psychostimulants in a treatment center (Kfar Izun) in Israel. The participants will undergo psychological evaluation before and during treatment and follow up at 4 months. Ten participants will undergo brain imaging of the dopamine receptor D2 in order to evaluate the effects of treatment on dopamine turnover in the brain. A control group of psychiatric in-patients undergoing treatment for psychiatric illness with be recruited from Geha Hospital in Israel. It is predicted that successful treatment of regular users of cannabis will be resulted in improvement in anxiety, depression and psychotic symptoms as well as in upregulation of dopamine turnover in participants that will undergo brain imaging.

DETAILED DESCRIPTION:
There is a significant number of cannabis and psychostimulant users that experience psychotic episodes and require psychiatric treatment. This study evaluates the effects of psychological and pharmacological treatment of regular users of cannabis and psychostimulants in a treatment center (Kfar Izun) in Israel. The participants will undergo psychological evaluation before and during treatment and follow up at 4 months. Ten participants will undergo brain imaging of the dopamine receptor D2 using [I123] IBZM in Single Photon Emitted Tomography (SPECT) before and after treatment in order to evaluate the effects of treatment on dopamine turnover in the brain. A control group of psychiatric in-patients undergoing treatment for psychiatric illness with be recruited from Geha Hospital in Israel.

ELIGIBILITY:
Inclusion Criteria:

* cannabis dependence with or without history of psychosis.

Exclusion Criteria:

* pregnant women
* under 18
* neurological damage
* HIV positive
* dependence on other drugs such as heroin
* cocaine or alcohol

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-10 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Questionnaire ratings of anxiety, depression and psychotic symptoms | 4 months
  Questionnaire measures of anxiety (Spielberger) Depression (BDI) and psychotic symptoms (PNAAS) will be used at baseline, during treatment and follow up at 4 months

SECONDARY OUTCOMES:
Dopamaine receptor D2 occupancy | At baseline and after 4 months
  Measures of dopamine receptor D2 occupancy using [I123] IBZM in Single Photon Emitted Tomography (IBZM) will be taken before and after treatment at 4 months.

CONTACTS AND LOCATIONS:
Overall Officials: Michal Roll, Ph.D, Study Director — Sourasky Medical Center
Locations (1):
- Sourasky Medical center, Tel Aviv, Israel